CLINICAL TRIAL: NCT02118480
Title: Improving Functional Disability and Cognition in Parkinson Disease: Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Deusto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSMC-001-UD
Record Dates: First submitted 2014-04-15; First posted 2014-04-21 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: PARKINSON DISEASE (Disorder)
Keywords: Parkinson disease, cognitive rehabilitation, REHACOP
MeSH Terms: conditions — Parkinson Disease | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cognitive remediation program: REHACOP (Experimental): Cognitive rehabilitation program (REHACOP) including intervention in: attention, memory, processing speed, language, executive functioning and social cognition during 3 months, 3 times per week
  Interventions: Other: cognitive remediation program: REHACOP
- Occupational Therapy (Active Comparator): The activities included drawing, reading the daily news and constructing using different materials (such as paper or wood) during 3 months, 3 times per week.
  Interventions: Other: Occupational Therapy

INTERVENTIONS:
Other: cognitive remediation program: REHACOP — Specifically, REHACOP group remediation with PD patients consisted of: Attention unit (4 weeks) training sustained, selective, alternant and divided attention; Memory unit (3 weeks) focusing on visual and verbal learning, recall and recognizing memory; Language unit (3 weeks) including grammar, syntax, vocabulary, verbal fluency, verbal comprehension, abstract language; Executive functions unit (2 weeks) training cognitive planning, proverbs, analogies; and Social cognition unit (1 week) exercising theory of mind, social reasoning and moral dilemmas.
  Arms: cognitive remediation program: REHACOP
Other: Occupational Therapy — The activities included drawing, reading the daily news and constructing using different materials (such as paper or wood). These activities were accomplished in a group format and with the same frequency as the implementation of REHACOP in the experimental group.
  Arms: Occupational Therapy

SUMMARY:
The study design was a parallel-group randomized trial with equal randomization. Recruitment and enrollment were conducted between June 2012 and January 2013. At base-line, clinical, cognitive and functional data was collected. Afterwards, the participants were randomly allocated to either the REHACOP group or the Control group. During 3 months the intervention with REHACOP program took place and at follow-up patients were again re-evaluated to evaluate the changes in clinical, cognitive and functional measures. Post-treatment assessment (finished by June 2013) was performed within the first week after completing the intervention.Optional enrollment in pre- post neuroimaging will also allow us to look at changes in the brain. Finally, longitudinal follow-up at 18 months with neuropsychological and neuroimaging assessements was also performed.

Objective: To examine the efficacy of an integrative cognitive training program (REHACOP) to improve cognition, clinical symptoms and functional disability of patients with Parkinson disease (PD).

DETAILED DESCRIPTION:
Assessment protocol:

- Cognitive Evaluation: The cognitive battery included assessments to evaluate processing speed, verbal learning and memory, visual learning and memory and executive functioning. All cognitive measures were converted into Z-scores based on the pooled PD group, and the sign of some measures was adjusted so that higher scores indicated better cognitive performance. All composite cognitive domains maintained satisfactory internal consistency. Processing Speed (Cronbach's α = 0.85) was quantified based on the Trail Making Test-A and Salthouse Letter Comparison Test. For verbal learning and memory (α = 0.88), learning and long-term recall performance on the Hopkins Verbal Learning Test (version 2 at baseline and 4 at post-treatment) were utilized. For visual learning and memory (α = 0.96), learning and long-term recall performance on the Brief Visual Memory Test (version 1 at baseline and 3 at post-treatment) were used (α = 0.96). Executive functioning (α = 0.78) was determined based on the Stroop test, using the word-color and interference scores.

Theory of mind (TOM). The strange stories test (Happé test) was administered to evaluate TOM. Four different stories (concerning double bluff, mistakes, persuasion and white lies) were administered at baseline and follow-up, and they were summed into a total TOM score with a possible range of 0 to 8. Higher scores indicate better TOM.

* Premorbid intelligence quotient and cognitive reserve. The Accentuation Reading Test (TAP), the Spanish version of the National Adult Reading Test (NART), was administered to calculate an estimation of each patient´s premorbid intelligence. The scale ranged from 0 to 30. Cognitive reserve was estimated using the Cognitive Reserve questionnaire. This 15-item multiple-choice questionnaire includes questions about education/culture, working activity, leisure and hobbies, physical activities and social activities. Higher scores indicate a better cognitive reserve, and the scale ranged from 0 to 26.
* Global cognitive status. The Mini-Mental State Examination (MMSE) was administered to obtain a general mental status score.
* Medication use. Medications, dosages and dose frequencies were used to calculate the levodopa-equivalent daily dose (mg/day) (LEDD).
* PD assessment. The Unified Parkinson's Disease Rating Scale and the Hoehn & Yahr scale were used for the assessment of the course and stage of the disease.
* Depressive symptoms. Geriatric Depression Scale (GDS-15) includes 15 items. Higher scores represent a higher degree of depression (range from 0 to 15).
* Neuropsychiatric symptoms. The NPI-Q was administered to evaluate neuropsychiatric symptoms. The test includes 10 items (delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, euphoria, apathy, disinhibition, irritability and aberrant motor behavior). These sub-scales were summed into a total score with a possible range of 0 to 120. Higher scores indicate more frequent and severe neuropsychiatric symptoms.
* Apathy. The Lille apathy rating scale consists of 33 items, including 9 sub-scales (everyday productivity, interests, taking initiative, novelty seeking/motivation, emotional responses, concern, social life and self-awareness). These sub-scales were summed into a total apathy score with a possible range of -36 to 36. Lower scores indicate less apathy.
* Functional disability. Functional disability was self administered using the World Health Organization Disability Assessment Schedule II (WHO-DAS II), short version (12 items).

Description of the intervention:

* REHACOP is a structured program using paper-pencil tasks and it is based on the principles of restoration, compensation and optimization with a gradually increasing level of cognitive effort and demand. REHACOP trains different cognitive domains, such as attention, memory, processing speed, language, executive functioning and social cognition. Additionally, the program includes one unit related to functional outcome: activities of daily living. REHACOP includes up to 300 different tasks hierarchically organized into at least three levels of difficulty and subtypes of abilities. Several tasks are timed, so processing speed is trained throughout various modules. Once a basic cognitive strategy has been trained and well acquired, the therapist transitions the program to the next level. The program format allows for either individual or group sessions (between 5 and 8 patients per group), although for the purpose of this study, group sessions were chosen. In this study, two psychologists conducted the REHACOP group attending 60-minute-long sessions 3 days per week at Parkinson Disease Association Biskay (ASPARBI) (two groups) or the Hospital of Galdakao (one group). Specifically, REHACOP group remediation with PD patients consisted of: Attention unit (4 weeks) training sustained, selective, alternant and divided attention; Memory unit (3 weeks) focusing on visual and verbal learning, recall and recognizing memory; Language unit (3 weeks) including grammar, syntax, vocabulary, verbal fluency, verbal comprehension, abstract language; Executive functions unit (2 weeks) training cognitive planning, proverbs, analogies; and Social cognition unit (1 week) exercising theory of mind, social reasoning and moral dilemmas.
* Occupational Activities: The Control group consisted of occupational group activities conducted by a psychologist at ASPARBI. The activities included drawing, reading the daily news and constructing using different materials (such as paper or wood). These activities were accomplished in a group format and with the same frequency as the implementation of REHACOP in the experimental group.

A subset of the sample will also complete a pre and post neuroimaging to evaluate changes in structural and functional brain activation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PD based on the United Kingdom PD Society Brain Bank (PDSBB) diagnostic criteria
* age 45-75 years
* either male or female
* Hoehn and Yahr disease stage 1-3 as evaluated by the neurologist

Exclusion Criteria:

* the presence of dementia as defined by the (DSM-IV-TR) Diagnostic and statistical manual of mental disorders IV Test Revised and the Movement Disorders Society specific clinical criteria for PD-dementia
* the presence of other neurological illness or injury (Traumatic Brain Injury, Multiple Sclerosis)
* unstable psychiatric disorders such as schizophrenia or major depression
* the presence of visual hallucinations as assessed by the Neuropsychiatric Inventory Questionnaire (NPI-Q)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in processing speed after receiving cognitive rehabilitation treatment | 3 months
Change in verbal memory performance after receiving cognitive remediation treatment | 3 months
Change in visual memory after receiving cognitive remediation treatment | 3 months
Change in executive functioning after receiving cognitive remediation treatment | 3 months
Change in theory of mind after receiving cognitive remediation treatment | 3 months

SECONDARY OUTCOMES:
Change in apathy after receiving cognitive remediation treatment | 3 months
Change in functional disability after receiving cognitive remediation treatment | 3 months
Change in depression after receiving cognitive remediation treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Naroa Ibarretxe-Bilbao, Doctor, Principal Investigator — University of Deusto
Locations (1):
- University of Deusto, Bilbao, Biskai, Spain

REFERENCES:
- [Derived] Pena J, Ibarretxe-Bilbao N, Garcia-Gorostiaga I, Gomez-Beldarrain MA, Diez-Cirarda M, Ojeda N. Improving functional disability and cognition in Parkinson disease: randomized controlled trial. Neurology. 2014 Dec 2;83(23):2167-74. doi: 10.1212/WNL.0000000000001043. Epub 2014 Oct 31. PMID 25361785